CLINICAL TRIAL: NCT05191667
Title: An Open-Label Multicenter Phase Ib Study of AN0025 in Combination With Chemoradiotherapy in Patients With Locally Advanced/Locally Recurrent Esophageal Cancer
Brief Title: AN0025 and Chemoradiotherapy Combination in Esophageal Cancer
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: The study is not stopped but the enrollment is suspended until a further decision from sponsor.
Sponsor: Adlai Nortye Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AN0025S0104
Record Dates: First submitted 2021-12-26; First posted 2022-01-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Paclitaxel; Carboplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with unresectable locally advanced/locally recurrent esophageal cancer (Experimental): Patients will receive AN0025 orally once daily (QD) and chemoradiotherapy followed by the maintenance of AN0025
  Interventions: Drug: AN0025

INTERVENTIONS:
Drug: AN0025 — 250 mg or 500 mg Q.D., oral administration
  Other Names: Paclitaxel; Carboplatin; Radiotherapy

SUMMARY:
This is an open-label, multicenter, phase Ib study to evaluate the safety, tolerability, and preliminary efficacy of AN0025 in combination with chemoradiotherapy (CRT) in patients with locally advanced/locally recurrent esophageal cancer.

DETAILED DESCRIPTION:
This study will enroll patients with unresectable locally advanced/locally recurrent esophageal cancer or esophagogastric junction cancer to assess the safety and tolerability of AN0025 at 250mg QD and 500mg QD combined with concurrent chemoradiotherapy to fix the MTD or RP2D. At RP2D level, another 20 patients with unresectable locally advanced/locally recurrent esophageal cancer or esophagogastric junction cancer will be enrolled at PR2D dose level to explore the preliminary efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with histologically- and/or cytologically-confirmed locally advanced/locally recurrent squamous cell carcinoma or adenocarcinoma of the esophagus or of the esophagogastric junction (EGJ).
2. Male or female, age≥18 years at the time of informed consent.
3. Have provided signed informed consent for the trial and are willing to comply with all aspects of the protocol

Exclusion Criteria:

1. With a history of another primary malignancy within the past 2 years, with the exception of basal or squamous cell skin cancer, or carcinoma in situ of the cervix or breast that has undergone potentially curative therapy.
2. Participants with known Hepatitis B or C infections, or known to be positive for Hepatitis B antigen (HBsAg)/ Hepatitis B virus (HBV) DNA or Hepatitis C antibody (HepC Ab)/ Hepatitis C virus (HCV) RNA. Active Hepatitis B is defined by a known positive HepB Ab result and known quantitative HBV DNA results greater than the lower limits of detection of the assay. Active Hepatitis C is defined by a known positive HepC Ab result and known quantitative HCV RNA results greater than the lower limits of detection of the assay.
3. Participants with known human immunodeficiency virus (HIV) infection (positive for HIV-1/2 antibody) or syphilis infection (positive for syphilis spiral antibody).
4. Major surgery or severe trauma within 4 weeks before the first dose of study drug. Note: If participant received major surgery, they must have recovered adequately from surgery and the toxicity and/or complications requiring the intervention prior to starting study treatment.
5. Have received prior systemic anti-cancer therapy including chemotherapy, target therapy, immunotherapy, anti-cancer traditional Chinese medicine, and other investigational oncology agents within 4 weeks or 5 half-lives, whichever is shorter. Participants who have entered the follow-up phase of an investigational study may participate as long as it has been at least 4 weeks (or 5 half-lives, whichever is shorter) after the last dose of the previous investigational agent.

   Note: Participants must have recovered from all AEs due to previous therapies to ≤ Grade 1 or returned to baseline. Participants with ≤ Grade 2 neuropathy or alopecia (per CTCAE v5.0) may be eligible.
6. Are currently participating in a study of an investigational device within 4 prior to the first dose of study treatment.
7. Have uncontrolled tumor-related pain.
8. Have a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.
9. Have a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Dose Limiting Toxicities (DLTs) | 4 weeks
  DLTs are defined as study drug-related toxicities graded using Common Terminology Criteria for Adverse events of the National Cancer Institute (NCI CTCAE) V5.0 occurring during DLT period (the first 4 weeks of AN0025 administration in combination with dCRT)

SECONDARY OUTCOMES:
Complete response rate (CRR) | 2 years
  The rate of patients with complete response in all tumor evaluable patients
Objective response rate (ORR) | 2 years
  The rate of patients with complete response and partial response in all tumor evaluable patients
Disease control rate (DCR) | 2 years
  The rate of patients with complete response, partial response and stable disease in all tumor evaluable patients
Progression-free survival (PFS) | 2 years
  The duration from the date of 1st dose to imageological progression or death, which earlier
Overall survival (OS) | 2 years
  The duration from the date of 1st dose to death

CONTACTS AND LOCATIONS:
Overall Officials: Jianming Xu, MD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Jianming Xu, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No